CLINICAL TRIAL: NCT03849378
Title: Effects of Sargassum Horneri Extract on Patients With Hypersensitivity
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Pusan National University Yangsan Hospital (Other)
Responsible Party: Principal Investigator, Sang Yeoup Lee, Professor, Pusan National University Yangsan Hospital
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: 02-2018-002
Record Dates: First submitted 2019-02-19; First posted 2019-02-21 (Actual); Last update posted 2022-04-26 (Actual); Status verified 2022-04

CONDITIONS: Skin Hypersensitivity

STUDY DESIGN:
Who Masked: Participant, Investigator
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Sargassum Horneri Extract group (Experimental): This group takes Sargassum Horneri Extract for 12 weeks.
  Interventions: Dietary Supplement: Sargassum Horneri Extract group
- Placebo group (Placebo Comparator): This group takes Placebo Extract for 12 weeks.
  Interventions: Dietary Supplement: Placebo group

INTERVENTIONS:
Dietary Supplement: Sargassum Horneri Extract group — This group takes 1,000 mg/day of Sargassum Horneri Extract for 12 weeks.
  Arms: Sargassum Horneri Extract group
Dietary Supplement: Placebo group — This group takes 1,000 mg/day of Placebo Extract for 12 weeks.
  Arms: Placebo group

SUMMARY:
The investigators conduct a randomized, double-blind, placebo-controlled study to investigate the effects of Sargassum Horneri Extract in patients with skin hypersensitivity for 12 weeks.

DETAILED DESCRIPTION:
Previous studies have indicated that Panax Ginseng C.A. Mey Extract may have the ability to improve liver function. Therefore, the investigators conduct a randomized, double-blind, placebo-controlled study to investigate the effects of the Sargassum Horneri Extract in patients with skin hypersensitivity for 12 weeks; the safety of the compound are also evaluate. The Investigators examine SCORAD(SCORing of Atopic Dermatitis) score, PGA (Patient Global assessment) score, IGA (Investigator Global assessment) score, total IgE, eosinophil counts, ECP, IL-4, IL-31, and TARC at baseline, as well as after 6 and 12 weeks of intervention. One hundred adults were administered either 1,000 mg of Sargassum Horneri Extract or a placebo each day for 12 weeks.

ELIGIBILITY:
Inclusion Criteria:

* Atopy by Hanifin & Rajka diagnostic criteria
* SCORAD < 40

Exclusion Criteria:

* Abnormal liver or renal function (i.e., serum aminotransferase activity > 3 times of upper limit of reference range and serum creatinine concentrations > 1.2 mg/dL)
* Diabetes (diagnosed clinically or fasting glucose level > 126 mg/dL)
* History of viral hepatitis or cancer
* Uncontrolled hypertension
* History of serious cardiac disease such as angina or myocardial infarction
* History of gastrectomy
* History of medication for psychiatric disease
* Administration of oriental medicine including herbs within the past 4 weeks

Ages: 12 Years to 50 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Child, Adult
Enrollment: 100 (Actual)
Dates: Start 2019-01-01 (Actual); Primary Completion 2022-02-14 (Actual); Study Completion 2022-02-28 (Actual)

PRIMARY OUTCOMES:
SCORing of Atopic Dermatitis (SCORAD) total score | Change from Baseline SCORAD total score at 3 months
  Change in SCORAD total score during 3 months

SECONDARY OUTCOMES:
Patient Global assessment (PGA) score | Change from Baseline PGA score at 3 months
  Change in PGA score during 3 months
Investigator Global assessment (IGA) score | Change from Baseline IGA score at 3 months
  Change in IGA score during 3 months
Total Immunoglobulin E (IgE) | Change from Baseline total IgE (IU/mL) level at 3 months
  Change in total IgE (IU/mL) level during 3 months
Eosinophil counts | Change from Baseline eosinophil counts (/uL) at 3 months
  Change in eosinophil counts (/uL) during 3 months
Eosinophil cationic protein (ECP) | Change from Baseline ECP (μg/L) level at 3 months
  Change in ECP (μg/L) level during 3 months
Interleukin-4 (IL-4) | Change from Baseline IL-4 (ng/mL) level at 3 months
  Change in IL-4 (ng/mL) level during 3 months
Interleukin-31 (IL-31) | Change from Baseline IL-31 (ng/mL) level at 3 months
  Change in IL-31 (ng/mL) level during 3 months
Thymus- and activation-regulated chemokine (TARC) | Change from Baseline TARC (pg/mL) level at 3 months
  Change in TARC (pg/mL) level during 3 months

CONTACTS AND LOCATIONS:
Overall Officials: Sang Yeoup Lee, MD, Principal Investigator — Pusan National University Yangsan Hospital
Locations (1):
- Pusan National University Yangsan Hospital, Yangsan, Gyeungsangnam-do, South Korea